CLINICAL TRIAL: NCT04015986
Title: Microbiota Directed Complementary Food (MDCF) Post-SAM MAM Trial
Brief Title: Community-based Clinical Trial With Microbiota Directed Complementary Foods (MDCFs) Made of Locally Available Food Ingredients for the Management of Children With Post-severe Acute Malnutrition Moderate Acute Malnutrition (Post-SAM MAM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR-18079
Record Dates: First submitted 2019-06-23; First posted 2019-07-11 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-01

CONDITIONS: Microbiota; Complementary Food; Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): MDCF-2 prototype with four complimentary food ingredients without powdered milk (rationale: lead with evidence from the recently completed pre-POC clinical trial of promoting growth promoting microbiota and positive effects on growth).
  Interventions: Dietary Supplement: Microbiota Directed Complementary Food-2
- Control arm (Active Comparator): Rice-lentil based RUSF (rationale: reference standard of care for post-SAM, MAM; based on knowledge of its effects on child growth and the gut microbiota)
  Interventions: Dietary Supplement: Ready to Use Supplementary Food

INTERVENTIONS:
Dietary Supplement: Microbiota Directed Complementary Food-2 — MDCF prototype with four complimentary food ingredients without powdered milk (rationale: lead with evidence from the recently completed pre-POC clinical trial of promoting growth promoting microbiota and positive effects on growth
  Other Names: MDCF-2
  Arms: Intervention arm
Dietary Supplement: Ready to Use Supplementary Food — Rice-lentil based RUSF (rationale: reference standard of care for post-SAM, MAM; based on knowledge of its effects on child growth and the gut microbiota)
  Other Names: RUSF
  Arms: Control arm

SUMMARY:
Background (brief):

1. Burden: A total of 52 million children under 5 are suffering from acute malnutrition globally, of whom 33 million suffer from moderate acute malnutrition (MAM). In Bangladesh, around 2 million children suffer from MAM. In absolute numbers, according to Bangladesh Demographic Health Survey 2014, 26%, 25% and 17% of children aged less than two years are stunted, underweight and wasted respectively.1
2. Knowledge gap: We have already demonstrated that children with acute malnutrition have immature gut microbiota that is partially corrected with treatment. Children with MAM have an increased risk of mortality, infections and impaired physical and cognitive development compared to well-nourished children. Although the global caseload of MAM is much greater than that of SAM, the condition has not received the same level of attention or priority. Through our previous and ongoing research we now know about the members of the gut microbiota that can promote growth in children and also about certain food ingredients that promote the proliferation of such beneficial microbiota. However, this knowledge needs to be applied on a large scale community-based clinical trial.
3. Relevance: The rationale for this study is to assess whether long-term administration of complementary food made of locally available food ingredients that can stimulate the proliferation of growth promoting gut microbiota (MDCF-2), as identified in our Pre-POC trial, is able to produce predictable changes in the microbiota of Bangladeshi children with Post-SAM MAM as well as in their nutritional status. We would now like to do a community-based clinical trial of this potential MDCF-2 in the management of children with Post-SAM MAM.

Hypothesis (if any): Complementary foods made of locally available food ingredients that stimulate the proliferation of growth promoting gut microbiota (MDCF-2) will improve clinical outcomes.

Objectives: To investigate the efficacy of complementary food made of locally available food ingredients that can stimulate the proliferation of growth promoting gut microbiota (Microbiota Directed Complementary Food: MDCF-2) in (i) promoting repair of microbiota immaturity (ii) promoting proliferation of beneficial bacteria (iii) improving both linear and ponderal growth in children with Post-SAM MAM (iv) improving the metabolomic profile of children with Post-SAM MAM

Methods: We will conduct a proof of concept (POC) clinical trial in 12-18 months old children with post-SAM MAM (Weight-for-Length Z-score, WLZ <-2 to -3) over the course of approximately two years. This study will be undertaken at Mirpur area of Dhaka city and in Kurigram. We will produce MDCF-2 at the icddr,b Food Processing Laboratory in sufficient quantities for the trial. This formulation is matched for energy density and micronutrient content of ready to use supplementary food (RUSF) used for MAM. It itself is not a ready-to-use food but is rather a cooked food made of locally available food ingredients (chickpea, green banana, peanut, soybean flour) which have been found to enhance growth promoting members of the gut microbiota in children. We will test MDCF-2 and the current RUSF standard of care for Post SAM MAM to see the effect on growth, proteomics and metabolomics of an intervention for 12 weeks, with a 4-week post-intervention phase.

Outcome measures/variables:

* Ponderal growth (rate of weight gain as the primary outcome variable), measured at different time points by anthropometry
* Linear growth, measured at different time points by anthropometry
* Proteomic profile, assayed by DNA aptamer based SOMAlogic scan
* Morbidity, assessed by daily records
* Change in microbiota-for-age Z score

Hypothesis to be tested:

Complementary food made of locally available food ingredients that can stimulate the proliferation of growth promoting gut microbiota (MDCF-2) will improve nutritional outcomes.

Specific Objectives To investigate the efficacy of complementary food made of locally available food ingredients that can stimulate the proliferation of growth promoting gut microbiota (Microbiota Directed Complementary Food: MDCF-2) in

(i) promoting repair of microbiota immaturity (ii) promoting proliferation of beneficial bacteria (iii) improving both linear and ponderal growth in children with Post-SAM MAM (iv) improving the metabolomic profile of children with Post-SAM MAM

DETAILED DESCRIPTION:
Background:

Moderate acute malnutrition (MAM), a major global health problem, is defined as wasting (i.e. weight-for-height between <-2 and -3 Z-scores of the WHO Child Growth Standards) and/or mid-upper-arm circumference (MUAC) greater or equal to 115 mm and less than 125 mm. According to the Global Nutrition Report 2017, 8% or 52 million under-five children were acutely malnourished globally in 2016 and stunting or chronic malnutrition affected 23% or 155 million children. Approximately one in 6 children under 5 years in South Asia suffered from MAM in 2013 (i.e. 17%). These children are at increased risk of severe acute malnutrition (SAM), and have a three times higher risk of mortality from common communicable diseases than the well-nourished peers. Bangladesh has one of the highest childhood malnutrition burdens in the world. According to Bangladesh Demographic Health Survey 2014, the prevalence of stunting in the country among under-five children is 36%, among them 12% suffer from severe stunting (LAZ <-3).1 Around 15% of children are wasted (weight-for-length, WLZ <-2); more than 2 million children suffer from MAM, while 3% or 450,000 children suffer from the deadly form of SAM. Malnutrition costs Bangladesh an estimated US $1 billion a year.

According to WHO recommendations, infants and children aged 6-59 months with MAM need to consume nutrient-dense foods to meet their extra needs for weight and height gain and functional recovery. Currently there are no evidence-informed recommendations on the composition of supplementary foods used to treat children with MAM. Interventions to address undernutrition should therefore include a strong component of MAM management. MAM prevention should be taken into consideration in food security and other development strategies as the situation becomes critical in populations where food insecurity is rampant. It is important therefore to develop interventions that depend upon locally available food ingredients which in small quantities are able to harness the beneficial power of the gut microbiota on infant and child growth.

One of the major factors limiting the impact of nutrition interventions is the inability of the malnourished children to increase their intake to meet increased metabolic demands. In collaborative studies between icddr,b and the Gordon Lab at Washington University in St. Louis during the Jumpstart Phase of the Breast Milk, Microbiota and Immunity (BMMI) Project, we applied Random Forests, to bacterial 16S rRNA (ribosomal RiboNucleic Acid ) datasets generated from monthly fecal samples obtained from a birth-cohort of children living in an urban slum of Dhaka, Bangladesh. These children exhibited consistently healthy growth (WLZ -0.32+0.98). Bacterial strains were identified whose proportional representation defines a healthy gut microbiota as it assembles during the first 2-3 postnatal years. In a randomized clinical trial at icddr,b of two therapeutic foods (imported ready-to-use therapeutic food [RUTF, Plumpy'Nut] versus locally prepared rice/lentil-based Khichuri and Halwa) in Bangladeshi children with severe acute malnutrition (SAM), it was observed that the microbiota immaturity is incompletely and only transiently improved, with children remaining markedly stunted and underweight throughout the follow-up period. Bangladeshi children with MAM also exhibited significant microbiota immaturity, although less severe than children with SAM. Microbiota immaturity thus serves as a potential biomarker to identify infants at risk for undernutrition and to monitor treatment and prevention strategies. In our previous study approved by the ERC (PR-09023), we compared the gut microbiota of healthy children living in slum of Mirpur with children hospitalized for the treatment of severe acute malnutrition. The microbiota was assessed by 16S Ribosomal RNA sequencing. We found that the gut microbiota of children with SAM lags chronologically behind microbiota of healthy children. For example, a two year old child with SAM may have the gut microbiota similar to that of a one year old healthy child. This is known as immaturity of the gut microbiota. We have developed two metrices to represent this gut immaturity - the relative microbiota maturity index and the microbiota-for-age Z score; SAM is associated with significant relative microbiota immaturity that is only partially ameliorated following nutritional interventions. .

We recently developed ready-to-use therapeutic foods using locally available food ingredients-rice, lentil, and chickpeas that are culturally relevant and acceptable. We found through a double-blind RCT (Randomized Controlled Trial ) that the Bangladeshi chickpea-based and rice-lentil-based RUTF (Ready To Use Therapeutic Food) we developed were as effective as the commercial peanut based-RUTF and well accepted by children with SAM. Through a combination of the above mentioned RCT and clinical translational studies conducted over the last 7-8 years, we have identified growth promoting age-discriminatory beneficial microbiota and locally available food ingredients that support proliferation of these beneficial microbiota. Besides, earlier studies done on gnotobiotic animals in Washington University Centre for Genome Science has led us to suggest that a combination of food ingredients (chickpea, soy flour, peanut and green banana) being informed by studies done in Dhaka will be worth studying with respect to the diet's impact on stimulating proliferation of growth-discriminatory microbiota as well as cost and sustainability.

Recently we successfully completed an IRB approved study, 'Pre-Proof of Concept clinical trials to optimize lead microbiota-directed complementary food (MDCF) prototypes for their ability to repair microbiota immaturity and establish their organoleptic acceptability' (PR-16099). The main objective of this pilot study was to demonstrate a Pre-proof of Concept that certain complementary foods would have a beneficial effect on young children suffering from MAM, by stimulating the proliferation of particular members of gut microbiota that are known for their growth promoting effects. In that pilot study we investigated Microbiota-for-age Z (MAZ) score as well as the impact of proliferation of good members of the gut microbiota on certain body systems. This study was designed to test the effects of three locally produced MDCF prototypes (MDCF-1, MDCF-2 and MDCF-3) and a locally produced rice-lentil-based RUSF. The results of the Pre POC pilot trial conclusively showed that one of the three MDCFs (namely MDCF-2) was associated with increased levels of certain amino acids that have a key role in development of long bones, development of the brain and increased production of IGF-1 (Insulin like Growth Factor-1) which are critical factors in the biology of child growth. Also it is effective in stimulating the growth of growth promoting members of the gut microbiota, for example Faecalibacterium prausnitzii. Based on the result of this Pre-POC pilot trial we now plan to do a larger clinical trial using the most promising MDCF-2 on the management of Post-SAM MAM children with the primary end point being linear growth.

Research Design and Methods We will conduct a clinical trial among 12-18 months old children with Post-SAM MAM (WLZ <-2 to -3) over the course of approximately two years. The trial will be conducted at Bauniabadh and RADDA MCH-FP clinic in Mirpur area of Dhaka city, and at the Special Nutrition Unit (SNU) run by Terre des Hommes (TdH) in Kurigram. The TdH SNU has been selected because we want to expedite the enrolment and we have a good track record of working there; the last efficacy trial we conducted on our local RUTFs was also done there partly. Children will be screened and enrolled through household survey by Field Research Assistants (FRAs) following pre-specified inclusion criteria. Fulfilling the enrolment criteria and upon receiving the consent for study participation from the parents or legal guardians, the children with the respective mother/caregiver will be enrolled and randomly assigned to one of the two arms according to computer-generated random numbers. The code of assigned type of diet will be kept in closed opaque envelopes for each individual, and will be opened only when the caregiver signs the consent form. This trial will not fall under any typical drug trial. However, if we are to consider this trial under any phase, then it would fall under phase II, because we have already done a pilot trial looking at the impact on microbiota-for-age Z score as well as adverse effects.

First of all, there will be the stabilization phase, which will be for 4-8 days, during that time each child will be managed as per WHO (World Health Organization) / icddr,b guidelines for the management of SAM. This includes programmed feeding, micronutrient supplementation, judicious rehydration, broad spectrum antibiotic treatment and prompt recognition and management of complications. Upon recovery from the stabilization phase nutritional rehabilitation will continue for approximately 2 weeks during which the icddr,b standard of care dietary protocol based upon the local diets Halwa and Khichuri will be served. Upon graduation from SAM to MAM (edema-free WLZ <-2), children will be randomly assigned to one of the two arms (Rice-lentil based RUSF and MDCF-2).

The post randomization nutritional rehabilitation component will have 3 phases. The first phase will involve onsite feeding of the diet twice daily for 1 month at the nutrition centres established in Mirpur and Kurigram. The second phase will entail feeding the children once at the nutrition center and once at home. During the third phase the children will be fed the diets twice daily at home. The children will be observed for 4 weeks in the post-intervention phase. During the entire study period, anthropometric data, food diversity data and samples (blood, stool, and urine) will be collected. We will collect weekly qualitative dietary intake data of over the last 24 hours by using Food Frequency Questionnaires during the dietary intervention for all study participants.

Randomization After the stabilization and nutritional rehabilitation phases when the children will reach to MAM state they will be randomly assigned to one of the two arms (Rice-lentil based RUSF and MDCF-2). The code of the assigned type of treatments will be kept in closed opaque envelopes until assigned to an enrolled child.

Arm 1- Rice-lentil based RUSF (rationale: reference standard of care for post-SAM, MAM; based on knowledge of its effects on child growth and the gut microbiota) Arm 2- MDCF-2 prototype with four complimentary food ingredients without powdered milk (rationale: lead with evidence from the recently completed pre-POC clinical trial of promoting growth promoting microbiota and positive effects on growth).

Recruitment, Screening and Consenting Children with SAM will be identified through direct observation and screening in icddr,b Dhaka Hospital, RADDA-MCH-FP Clinic in Mirpur, the SNU of TdH in Kurigram, as well as through screening in the communities in Mirpur and Sadar, Ulipur and Chilmari Upazilas of Kurigram district. Those who require stabilization care will be admitted in the facilities mentioned above where the standard of care for the acute phase treatment of SAM will be provided. In brief; this stabilization care is based upon programmed feeding, micronutrient supplementation, judicious rehydration, broad spectrum antibiotic treatment and prompt recognition and management of complications. They will subsequently be treated with the standard of care dietary protocol for nutritional rehabilitation. Upon graduation into MAM, parents of children who meet the MAM criteria for post-SAM MAM trial will be approached about enrolment into the study. A trained Field Research Assistant (FRA) will explain the study in detail, answer any questions from the parent(s), and invite the parent(s) to enrol the child in the study.

At the beginning of the study, information will be sought on the demographic characteristics and FRAs will record the children's weight using a digital scale with 2 g precision (Seca, model 728, Germany), length (using infantometer, Seca, model 416, Germany), and mid-upper-arm circumference to the nearest mm (using a non-stretch insertion tape). Anthropometrics will be done according to the standard procedures. Study participants will be asked to come to the designated nutrition center for nutritional therapy to ensure intake of the MDCF/RUSF. They will be provided with a phone number to reach the clinic staff, and a member of the staff may visit a family's household for directly observed nutritional therapy with prior arrangement if needed. The programmed feeding of the MDCF-2 or RUSF for three months after nutritional rehabilitation is illustrated in the figure.

Preparation of MDCF-2 and RUSF:

Based on compatible combinations of complementary food ingredients identified in the Pre-POC study mentioned above, we will prepare MDCF-2 as well as RUSF at the icddr,b Food Processing facility in Mirpur and in Kurigram in sufficient quantities for the clinical study. The two diets will be matched in energy density and micronutrient content. The energy density of MDCF-2 is targeted at 125 kcal/25 g (per serving), and caloric distribution is targeted to be 45-50 percent from fat and 8-10 percent from protein. The two servings of MDCF-2 or RUSF will provide 250 Kcal and the necessary micronutrients in addition to providing the substrate for the beneficial microbiota proliferation. The servings are meant to be a top up to the usual diet received by these children at home. Mothers/primary caregivers will be advised to maintain their child's current dietary and breastfeeding practices.

Experiments in development of the MDCF-2 prototypes and assessment of the organoleptic properties have been done in the Pre-POC clinical trial.

Food will be prepared everyday to ensure that no unexpected contamination and nutrient losses occur during preparation. Although raw food ingredients will be very carefully procured from the local market and stored in reasonable quantities, we will prepare, dispense, and feed the children the same day the MDCF-2 and RUSF are prepared.

After receiving the raw materials (rice/lentil/chickpea) we will take out the foreign materials/grains or seeds (if there is any) those can be discarded, and then in an open pan the raw materials will be roasted. We will maintain the temperature at 120-130°C for roasting. Usually it takes 8-10 minutes for roasting 100g of each raw material. Continuous stirring is essential to ensure roasting of single seeds/grains. After completion of roasting we will keep it aside for cooling and then we will grind. We will take the powder and strain it using a strainer. After straining for 4 to 5 times, we will take the fine powder for mixing with the other ingredients (milk powder/oil). We will also grind the sugar and the fine powder will be used for mixing. Finally we will add the pre-weighed premix powder. The processing of whole green banana is different from the other ingredients. Green banana with skin will be placed in a deep pan in boiling water (100°C-110°C) and boiled for about 17-20 minutes until they are cooked and tender. The skin of the green banana will be peeled off and the edible white part would be taken and grated into small pieces. Then they will be taken in a pot and allowed to cool. We will smash the small pieces of banana with spoon/hand crusher. The weights of all other ingredients will be recorded. Potential recipes will be produced in small batches by mixing all ingredients in an electric blender. Preparation of food under different steps, that is, roasting, particle size reduction, homogeneous blending, and supplying to the nutrition centres will be monitored by icddr,b investigators. Food will be prepared everyday to ensure that no unexpected contamination and nutrient losses occur during preparation. Although raw food ingredients will be very carefully procured from the local market and stored in reasonable quantities, we will prepare, dispense, and feed the children the same day the MDCF and RUSF are prepared.

Feeding sessions:

The children and mothers/caregivers will be requested to come to the nutrition centers established at the sites preferably between 9-11 am and 3-5 pm every day for the first month. The mothers will be requested not to give any food and breast milk in the 2 hours preceding the observed meal time. The child will be offered 25 grams of MDCF-2 or RUSF per serving as decided by randomization. The mothers will be asked to spoon feed the pre-weighed diets to their children until s/he refuses to eat, as described below. After a two-minute pause, the same diet will be offered a second time until s/he refuses again. After a second two-minute pause, the diet will be offered a third time until refused again. After this third refusal, the feeding episode will be considered as 'terminated'. The duration of the feeding (excluding the intervening 'rest periods') will be recorded by stopwatch, and the total duration of the feeding will be noted. This feeding episode will last for maximum 60 minutes. Measured volumes of plain water will also be given and the amount of water taken during this meal period of 60 minutes will be measured. The feeding episode will take place under the direct supervision of trained study personnel. Children will be considered as refusing further intake if they move their head away from the food, cry, clamp the mouth or clinch the teeth, or become agitated, spit out the food or refuse to swallow. The amount of MDCF-2/RUSF actually ingested will be calculated by subtracting the left over from the offered amount, or by asking the mother when fed at home. The enrolled children will be monitored daily by Field Research Assistants for any possible side effects/adverse events (e.g. rash, urticaria due to food allergy or any significant changes in clinical status) for a week. If any side effects/adverse events are observed, they will be treated according to standard of care. A standardized production procedure will be followed to control the quality of RUSF and MDCF-2. Every child will be offered 25gm of the diet twice daily at the feeding center for the first 4 weeks. In the following month, the child will be offered 25gm of the diet at the feeding center and additional 25gm will be provided in a clean container to feed at home. In the third month, two separate containers containing 25gm diet will be provided every day to each enrolled child at participant's home. Feeding information will be collected from mothers and amount consumed will be measured from the left outs. Food will be kept in sterile containers and at room temperature in between the feeding session. Quality of the food will be ensured by having samples of the prepared foods tested for microbes and moulds every 2 months at icddr,b. Samples selected for testing will include food stored for 2 and 6 hours after cooking. The samples will also be tested for Aflatoxin every six months at SGS Laboratories, Delhi.

In this study nutritional status will be assessed through anthropometry, comparing with WHO growth reference standards. At the beginning of the study, information will be sought on the demographic characteristics (families' wealth, standard of housing, family structure and parental characteristics etc.), and FRAs will record the children's weight using a digital scale with 2g precision (Seca, model 728, Germany), length (using infantometer, Seca, model 416, Germany), and mid upper-arm circumference to the nearest mm (using a non-stretch insertion tape). Anthropometrics will be done according to the standard procedures and all measurements will be taken thrice and the average value will be recorded.

Fecal sample collection In acute phase of stabilization fecal samples will be collected every alternative day. During the rehabilitation phase, weekly fecal samples (1-2g) will be collected within 30 minutes of production (at home and transported back to the icddr,b) using the Nitrogen dry shipper specimen collection SOP (Standard Operating Procedure) used in the recent Pre-POC clinical trial (Appendix-A). Specimens will be stored at -80◦C before being sent to the Gordon Lab at the end of each study for analysis of microbiota maturity (measured before, during and after cessation of treatment with MDCF-2 and RUSF) and PCR-based assessment of enteropathogen burden in fecal samples (measured before and after MDCF-2 treatment). A total of 12 fecal samples will be collected from each child at different time points during whole study period. Assuming 62 study participants / arm, a total of 1488 fecal specimens will be collected in this study. Along with that 2 gm of fecal sample will be collected from the mothers at the beginning of stabilization phase.

Urine sample collection A total of 7 urine samples (2 ml each) will be collected from each child at different time points during the whole study period. Assuming 62 study participants / arm, a total of 868 urine samples will be collected in this study. Along with that 5 ml of urine samples will be collected from the mothers at the beginning of stabilization phase.

Blood sample collection A total of 4 blood samples (2 ml each) will be collected at different time points during the whole study period. Each will be collected from every child at the beginning of stabilization phase, prior to intervention; end of first month of intervention and just after the intervention is complete.

Assuming 62 study participants / arm, a total of 496 plasma samples will be collected in this study. Along with that, 5 ml of blood samples will be collected from the mothers at the beginning of stabilization phase.

Maternal nutritional status is associated with child nutritional status, as shown through the results of our eight country MAL-ED study. In addition, antenatal and maternal factors were early determinants of lower length-for-age, and their contribution remained important throughout the first 24 months of life. As such, we will record maternal height and weight. In order to understand the biological state of nutrition of the mother, enrolment samples of stool, blood and urine will be asked of the mother. These samples will be analyzed for gut microbiota, and proteomics, and the results correlated with those of the enrolled children.

Anthropometry The age of the child will be verified against documentation (birth certificate or immunization card, if available) or caregiver's report of the child's birth date. Length will be measured by a infantometer sensitive to 0.1 cm. Body weight will be measured by a balance sensitive to 2g (SECA 7281321009, Hamburg, Germany). Length-for-age (LAZ), weight-for-length (WLZ) and weight-for-Age (WAZ) Z-scores will be calculated following the Multicentre Growth Reference Study (MGRS) WHO growth standards. Edema will be examined by pressing the upper side of both feet for 3 seconds. Mid-upper arm circumference (MUAC) will be measured using TALC MUAC tape (UK). Regular standardization of the measuring equipments will be done using standards everyday by trained field research assistant.

Analyses of plasma and fecal samples Plasma samples collected from this trial will be sent to Dr Jeffrey Gordon's lab in the Center for Genome Sciences and Systems Biology at Washington University in St. Louis. Advanced mass spectroscopic- and immunoassay-based methods will be used to obtain new knowledge about the role of gut microbiota immaturity and the effects of attempting acute repair of this immaturity with lead microbiota-directed complementary food (MDCF-2) on biomarkers and mediators of healthy growth. Comparisons will be made with the control group (i.e., those consuming reference RUSF standard). Targeted Ultra Performance Liquid Chromatography-Mass Spectrometry (UPLC-MS) and Gas Chromatography-Mass Spectrometry (GC-MS) will be used to profile analytes of specific interest in plasma and/or fecal samples including bile acids and short chain fatty acids (SCFAs); markers of mitochondrial function (e.g., β-hydroxybutyrate, acylcarnitines/acylCoAs, TCA cycle intermediates); amino acids in serum plus fecal samples [branch chain amino acids, tryptophan and tryptophan metabolites related to growth and inflammatory status, including those produced by bacterial tryptophan metabolism (e.g. indole acetic acid derivatives)]. In addition, key mediators/biomarkers of linear growth (e.g., growth hormone and IGF-1), energy utilization (insulin, leptin), and bone biology [IL-6 (interleukin-6), osteoprotegerin, the C-terminal peptide of type I collagen (CTX, a marker of osteoclast activity/bone resorption), and the amino-terminal propeptide of Type 1 procollagen (P1NP, a marker of osteoblast activity/bone formation)], and systemic inflammation (CRP, AGP) will be quantified using established ELISA/Luminex assays. Proteins in blood will be identified using the SOMAlogic scan that permits identification of more than 1300 different proteins. The proteomic study done on plasma samples from children with SAM in our previous Pre-POC trial done in Dhaka has already demonstrated a number of significant and clinically relevant associations between certain proteins and clinical phenotypes using the SOMAlogic scan.

Information gathered will be used to select human fecal samples for transplantation into germ-free animals; these animals, who will be fed the diets of their human microbiota donors, will be used to further characterize the mechanisms that link MDCF-2 prototypes, the gut microbiota, and host physiology/metabolism. In addition, these plasma and fecal biomarkers will be used to determine that MDCF-2 promotes repair of microbiota immaturity and improves biological state in children.

Sample Size Calculation In the pre-POC trial of different MDCFs, the baseline weight-for-length Z score of children who received MDCF2 (Microbiota Directed Complementary Food 2) was -2.2 and after one month of supplementation was -1.7. If we consider the WLZ -2 at baseline and -1.7 at end line, pooled SD (standard deviation) as 0.53 then the sample size is 49 in each arm at 80% power and 5% level of significance. With 20% attrition 62 children will be required to be enrolled in each arm. Therefore, for this trial, 62 children will receive MDCF-2 and 62 children Rice-lentil RUSF.

Data Analysis:

The two groups of children with Post SAM-MAM will be compared at baseline and at different time points as shown in the illustration on trial design. The clinical outcome variables for comparison will include rate of weight gain, anthropometric indices, and morbidity. All analytes mentioned in the section 'Analyses of plasma and fecal samples' will be compared between MDCF-2 and RUSF groups.

Ethical Assurance for Protection of Human rights The study has been started after obtaining IRB (Institutional Review Board ) approval by the icddr,b Research Review Committee and Ethical Review Committee. Before enrolment in the study, informed written consent are being taken from the legal guardian of the study participants. Personal identifications taken during enrolment and other study procedures are being kept under lock and key.

Expected risks/adverse events for this protocol are those related to blood sample collection, fecal sample collection and feeding of microbiota directed complementary food. None of these qualify as a serious adverse event (SAE). Expected Adverse Events (EAEs) related to blood draw are as follows:

* discomfort
* pain
* introduction of infection
* bleeding
* fainting or bruising

  * Precaution will be taken to avoid introduction of infection by disinfecting the site of venipuncture and using sterile equipment
  * The risk of bleeding and bruising will be minimized by immediate application of pressure after venipuncture
  * The participant (child) will be in the sitting or supine position during blood draws to avoid injuries from fainting

All possible adverse events will be treated appropriately. These will include:

* Vomiting
* Diarrhoea
* Skin rash
* Urticaria from food allergy
* Abdominal distension
* Pain abdomen Assessment of Adverse Events Both serious and non-serious adverse events will be assessed for severity; relationship to study participation; actions taken; and outcomes. All SAEs must be reported to the ERC (Ethical Review Committee) of icddr,b within 24 hours of the site's awareness of the event that will in turn be distributed to the sponsor. This will be done by direct telephone communication, fax or e-mail.

icddr,b IRB recommended guidelines would be followed for grading the adverse events, if any that take place.

Severity:

1. Mild
2. Moderate
3. Severe

Relationship to Study participation:

1. Definitely related:Clear cut temporal association, no other possible cause
2. Possibly related:Less clear cut temporal association, other causes possible
3. Unrelated: Independent of study, evidence exists that event is definitely related to another etiology

Actions:

None Remedial therapy (more than one dose of medicine required) Permanently discontinued from study participation Hospitalization Other

Outcomes:

Resolved Continuing Unknown Collaborative Arrangements This project is a collaborative effort between the investigators at the Washington University School of Medicine and the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b). The clinical works, field activities will be undertaken in Dhaka and Kurigram, Bangladesh, under the direct supervision of the Principal Investigator whereas the laboratory analyses will be conducted at the Gordon Lab at Washington University in St. Louis. All research units and the collaborating investigators have long histories of international collaborations. All investigators have communicated during development of this project and are committed to its successful implementation.

Facilities Available icddr,b has a well-equipped Food Processing Lab that will facilitate experiments on the diet recipes. We have ongoing studies in the Baoniabad area in Mirpur. A number of project offices are located there. More importantly, we have an excellent rapport with the community. The Terre des Hommes that runs the SNU in Kurigram where a part of the trial will be conducted. In the past we helped in the development of the SNU and have performed studies there. The SNU has a great reputation in the community.

Center for Genome Sciences, Washington University in St. Louis:

The stool samples will be aliquoted at icddr,b. Stool samples will be sent to Prof Jeffery Gordon's Lab in St Louis for the high throughput 16S ribosomal RNA gene sequencing. The presence/abundances of a broad range of enteropathogens in stool samples before and after MDCF-2 treatment will be determined using a PCR (Polymerase Chain Reaction)-based assay. Stool samples may also be used to culture constituent bacterial strains for use in future studies in gnotobiotic mice in the Gordon Lab. It is pertinent to mention here that the assays and equipment to carry out those are currently available only in a few labs in the world, including the one at St Louis. The Center is home to an interdisciplinary, multi-departmental, multi-generational team of investigators from multiple schools that focus on comparative genomics, statistical genomics, and systems biology It serves as 'proving ground' for developing new strategies for educating students and faculty who wish to work at the interface of the biological, physical, computational and engineering sciences.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s) willing to sign consent form; the informed consent document will explicitly request permission to use the collected fecal samples for future studies, including but not limited to culturing component bacterial strains
* Child age 12-18 months
* WLZ between <-2 and -3 without bilateral pedal edema at the time of randomization
* Parent(s) willing to bring the child to the feeding centre twice daily for 4 weeks for nutritional therapy, once daily for next 4 weeks and administer the feeds provided by study staff once daily at home for 4 weeks and twice daily for next 4 weeks.

Exclusion Criteria

* Medical conditions: Children with tuberculosis (diagnosis based on WHO 2014 guidelines which have been incorporated in the national TB control guidelines of Bangladesh). The guidelines depend upon the following five diagnostic principles (three out of five should be positive): 1. Specific symptoms of TB, 2. Specific signs, 3. Chest X-ray, 4. Mantoux test, and 5. History of contact,[9] or any congenital/acquired disorder affecting growth i.e. known case of trisomy-21 or cerebral palsy; children on an exclusion diet for the treatment of persistent diarrhea; having known history of soy, peanut or milk protein allergy- Severe anemia (<8mg/dl), will be assessed by Hemocue (Model no. Hemocue Hb 301)
* Failure to obtain informed written consent from parents or caretakers

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Ponderal growth | At the enrollment (day1), every day during acute phase and nutritional rehabilitation phase, every 15 days during the 3 months of intervention phase and at the end of 1 month of follow up phase by anthropometry
  Rate of weight gain of the enrolled participants
Change in Liner growth (LAZ) | At the enrollment (day1), every week during the acute phase and nutritional rehabilitation phase, every 15 days during the 3 months of intervention phase and at the end of 1 month of follow up phase by anthropometry
  Rate of skeletal human growth
Change in Proteomic profile | A total of 4 plasma samples will be collected, at enrollment, prior to 3 months of intervention, end of first month of intervention and just after the completion of intervention.
  Information about all proteins that are made in blood, other body fluids, or tissues, at certain times.It will be assayed by Somalogic scan
Change in Morbidity | Data will be collected every day from enrollment, during the acute and rehabilitation phase, 3 months of intervention phase and once at the end of 1 month of follow up phase.
  Refers to having a disease or a symptom of disease. It will be assessed by taking morbidity data
Change in Microbiota-for-Age Z (MAZ) score | At enrollment, every alternative day during the stabilization phase, once during the nutritional rehabilitation phase, weekly during the first month of intervention, at the end of 2nd and 3rd months of intervention & at the end of 1 month of follow up.
  bacterial species whose proportional representation define a healthy gut microbiota as it assembles during the first two postnatal years of life. 'microbiota-for-age Z-score' compares development of a child's fecal microbiota relative to healthy children of similar chronologic age.

CONTACTS AND LOCATIONS:
Overall Officials: Tahmeed Ahmed, PhD, MBBS, Principal Investigator — Senior Director, Nutrition & Clinical Services Division, icddr,b; Munirul Islam, PhD, MBBS, Study Chair — Senior Scientist, Nutrition and Clinical Services Division, icddr,b; Sayeeda Haque, MPH, MBBS, Study Chair — Associate scientist, Nutrition and Clinical Services Division, icddr,b; Ishita Mostafa, MPH, MBBS, Study Chair — Research Investigator, Nutrition and Clinical Services Division, icddr,b; Imteaz Mahmud, MBBS, Study Chair — Research Fellow, Nutrition and Clinical Services Division, icddr,b; Nurun Nahar Naila, MPH, MBBS, Study Chair — Assistant Scientist, Nutrition and Clinical Services Division, icddr,b; Mustafa Mahfuz, MPH, MBBS, Study Chair — Associate scientist, Nutrition & Clinical Services Division, icddr,b
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mostafa I, Nahar NN, Islam MM, Huq S, Mustafa M, Barratt M, Gordon JI, Ahmed T. Proof-of-concept study of the efficacy of a microbiota-directed complementary food formulation (MDCF) for treating moderate acute malnutrition. BMC Public Health. 2020 Feb 17;20(1):242. doi: 10.1186/s12889-020-8330-8. PMID 32066412